CLINICAL TRIAL: NCT01061125
Title: Implantable Loop Recorders in Post-AF Ablation: RPAF-A
Brief Title: Implantable Loop Recorders in Post-atrial Fibrillation (AF) Ablation: RPAF-A
Acronym: RPAF-A
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Walid Saliba, MD, The Cleveland Clinic
Other Study IDs: 09-212
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; implantable loop recorder; TTM
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unblinded: Transtelephonic (TTM) monitoring weekly for 5 months Holter monitor recording at 4 months and at 12 months Implantable Loop Recorder (ILR) weekly reports
  Interventions: Other: TTM and Holter monitor
- Blinded: TTM and Holter Monitor conventional follow up Implantable Loop Recorder (ILR) unblinded at 5 months
  Interventions: Other: TTM and Holter monitor

INTERVENTIONS:
Other: TTM and Holter monitor — Standard of care visits recordings reviewed during clinical visits
  Other Names: Transtelephonic monitoring

SUMMARY:
This is a randomized pilot study, of post pulmonary vein isolation (PVI) patients to determine the clinical utility of the Implantable Loop Recorder. These type of patients either are monitored with weekly transtelephonic monitoring (TTM) or implantable loop recorder (ILR). The Medtronic Reveal XT loop recorder will be implanted at the time of the PVI or at the 3-4 month PVI follow-up visit and patient care will be managed based on randomization to a blinded or unblinded group. Outcome measures will be compared to aid in decision making regarding anticoagulation and overall post ablation clinical management.

DETAILED DESCRIPTION:
This is a randomized pilot study, of post pulmonary vein isolation (PVI) patients to determine the clinical utility of the Implantable Loop Recorder. The Medtronic Reveal XT implantable Loop Recorder is a market released device indicated for patients with clinical syndromes or situations at increased risk of cardiac arrhythmias, and patients who experience transient symptoms that may suggest a cardiac arrhythmia. These type of patients either are monitored with weekly transtelephonic monitoring (TTM) or implantable loop recorder (ILR). Neither approach has been shown to be superior. As both approaches are currently being performed based on physician preference, the investigators propose to study and compare both approaches in a randomized fashion for evidence based practice. The Medtronic Reveal XT loop recorder will be implanted at the time of the PVI or at the 3-4 month PVI follow-up visit and patient care will be managed based on randomization to a blinded or unblinded group. Outcome measures will be compared to aid in decision making regarding anticoagulation and overall post ablation clinical management.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation
* Chads score > or equal to 1

Exclusion Criteria:

* contraindication for ILR
* life expectancy less an 12 months
* pregnant women
* existing cardiac rhythm management (CRM) device

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for atrial fibrillation ablation
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
AF Burden Conventional Follow up | Weekly for five months
  TTM and Holter Monitor Transmissions

CONTACTS AND LOCATIONS:
Overall Officials: Walid Saliba, MD, Principal Investigator — The Cleveland Clinic; Oussama Wazni, MD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No